CLINICAL TRIAL: NCT05782179
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Safety, Tolerability and Immunogenicity of Three Doses of Group B Streptococcus Vaccine (GBS NN/NN2 With Alhydrogel®) in Elderly Participants Aged 55 to 75
Brief Title: Study to Evaluate the Safety, Tolerability and Immunogenicity of Three Doses of GBS Vaccine in Elderly Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Minervax ApS (Other)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MVX0006; 2022-003681-20 (EudraCT Number)
Record Dates: First submitted 2023-02-23; First posted 2023-03-23 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Group B Streptococcal Infections
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1 - Active (Experimental): Cohort 1 (30 healthy older adult) will receive three injections, each consisting of 50 μg of GBS-NN and 50 μg of GBS NN2 bound to aluminium hydroxide in a 4:1 ratio (investigational medicinal product or placebo).
  Interventions: Biological: GBS-NN/NN2
- Cohort 1 - Placebo (Placebo Comparator): Cohort 1 (30 healthy older adult) will receive three injections, each consisting of 50 μg of GBS-NN and 50 μg of GBS NN2 bound to aluminium hydroxide in a 4:1 ratio (investigational medicinal product or placebo).
  Interventions: Biological: Placebo
- Cohort 2 - Active (Experimental): Cohort 2 (30 healthy older adult) will receive three injections, each consisting of 125 μg of GBS-NN and 125 μg of GBS NN2 bound to aluminium hydroxide in a 4:1 ratio (investigational medicinal product or placebo).
  Interventions: Biological: GBS-NN/NN2
- Cohort 2 - Placebo (Placebo Comparator): Cohort 2 (30 healthy older adult) will receive three injections, each consisting of 125 μg of GBS-NN and 125 μg of GBS NN2 bound to aluminium hydroxide in a 4:1 ratio (investigational medicinal product or placebo).
  Interventions: Biological: Placebo
- Cohort 3 - Active (Experimental): Cohort 3 (15 obese and/or diabetic older adults) will receive three injections, each consisting of 50 μg of GBS-NN and 50 μg of GBS NN2 bound to aluminium hydroxide in a 4:1 ratio (investigational medicinal product or placebo).
  Interventions: Biological: GBS-NN/NN2
- Cohort 3 - Placebo (Placebo Comparator): Cohort 3 (15 obese and/or diabetic older adults) will receive three injections, each consisting of 50 μg of GBS-NN and 50 μg of GBS NN2 bound to aluminium hydroxide in a 4:1 ratio (investigational medicinal product or placebo).
  Interventions: Biological: Placebo
- Cohort 4 - Active (Experimental): Cohort 4 (15 obese and/or diabetic older adults) will receive three injections, each consisting of 125 μg of GBS-NN and 125 μg of GBS NN2 bound to aluminium hydroxide in a 4:1 ratio (investigational medicinal product or placebo).
  Interventions: Biological: GBS-NN/NN2
- Cohort 4 - Placebo (Placebo Comparator): Cohort 4 (15 obese and/or diabetic older adults) will receive three injections, each consisting of 125 μg of GBS-NN and 125 μg of GBS NN2 bound to aluminium hydroxide in a 4:1 ratio (investigational medicinal product or placebo).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GBS-NN/NN2 — GBS-NN/NN2 bound to alhydrogel as an adjuvant
  Arms: Cohort 1 - Active; Cohort 2 - Active; Cohort 3 - Active; Cohort 4 - Active
Biological: Placebo — Normal Saline 0.9 %
  Arms: Cohort 1 - Placebo; Cohort 2 - Placebo; Cohort 3 - Placebo; Cohort 4 - Placebo

SUMMARY:
The study is a randomised, double-blind, placebo-controlled, parallel group study to evaluate the safety, tolerability and immunogenicity of three doses of GBS NN/NN2 with Alhydrogel® (Recombinant protein vaccine against Group B Streptococcus) in elderly participants aged 55 to 75.Participants will be followed up to 6 months after last vaccination.

DETAILED DESCRIPTION:
Sixty (60) healthy older adult participants aged 55 to 75 years will be randomised in two cohorts; 30 obese and/or diabetic participants aged 55 to 75 years will be randomised in two cohorts.

Participants will be involved in the study for approximately one year including screening and safety follow-up.

Eligible participants will be administered a dose of GBS-NN/NN2 or placebo on three occasions: the first dose will be administered on Day 1, followed by the second and third doses 4 and 24 weeks later, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 55 to 75 years.
2. Body mass index (BMI) ≥18 and ≤30 kg/m2 for healthy participants, ≥ 30 to ≤45 kg/m2 for obese participants and ≥18 to ≤45 kg/m2 for type 2 diabetic participants.
3. Able to voluntarily provide written informed consent to participate in the study.
4. Female participants must be post-menopausal.
5. Participants capable and willing to follow trial schedule and procedures.

Exclusion Criteria:

1. Participants who have received a GBS vaccine previously.
2. Participants with history or presence of significant (as evaluated by the investigator) cardiovascular disease, pulmonary, hepatic, gallbladder or biliary tract, renal, haematological, gastrointestinal, endocrine, immunologic, dermatological, neurological, psychiatric, autoimmune disease or current infection.

   NOTE: Patients with type 2 diabetes are to be recruited for Cohort 3 and Cohort 4.
3. Laboratory values at screening which are deemed by the investigator to be clinically significantly abnormal.
4. Current or history of drug or alcohol abuse per investigator judgement.
5. Positive for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
6. Participants currently participating in a clinical trial.
7. Participants receiving an investigational drug, vaccine or device during the 90 days preceding the initial dose in this study.
8. Any significant illness during the 4 weeks preceding the vaccination visit, per investigator judgement.
9. Participants with a history of severe allergic reactions after previous vaccination.
10. Participants who have received any vaccine within 30 days of first IMP administration, or who are planning to receive any vaccine (eg, travel vaccines) up to 30 days after each vaccination.

    NOTE: Exceptions could be made for emergency vaccinations (eg, tetanus) or vaccination campaigns (eg, SARS, CoV-2 or influenza) which will be permitted not less than 7 days before or after study vaccination.
11. Participants receiving immunosuppressive therapy or immunoglobulins in the 6 months prior to screening.
12. Participants within a 7-day period after an acute infection in the 7 days preceding vaccination, as per investigator judgement, or with fever (oral temperature >37.9°C) in the 72 hours preceding vaccination.
13. Participants who have received antipyretics/analgesics treatment within 72 hours prior to dosing.
14. Participants on chronic medications that are likely to affect the assessments specified in the protocol (eg, anticoagulant therapy, systemic steroids).

    NOTE: Chronic medications such as antihypertensives, bronchodilators, statins that do not affect the immune system, will be permitted and allowed to continue during the study at the discretion of the investigator. Treatment for diabetes will be continued as required for the diabetic participants recruited. Non-steroidal anti-inflammatory drugs or paracetamol will be permitted for the treatment of headache or other symptoms during the study. Use of over the counter (OTC) vitamins and dietary supplements is allowed.
15. Participants with skin defects and/or tattoos at the proposed site of vaccine administration.
16. Donation of blood or blood products within 90 days prior to first study vaccination.
17. Participants who, in the opinion of the Investigator, are unsuitable for participation in the study.
18. Involvement in the planning and/or conduct of the study (applies to both Sponsor personnel and/or personnel at the study centre or Clinical Research Organisation [CRO]).

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Kitson, Study Director — gkitson@propharmapartners.uk.com
Locations (1):
- University Hospital Ghent - Centrum voor Vaccinologie (CEVAC) department, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 90 participants were enrolled and randomised.
Groups:
- Healthy Older Adult : GBS-NN/NN2 50 µg: Healthy older adult received three injections, each consisting of 50 μg of GBS-NN and 50 μg of GBS NN2 bound to aluminium hydroxide.
  GBS-NN/NN2: GBS-NN/NN2 bound to alhydrogel as an adjuvant
- Healthy Older Adult : GBS-NN/NN2 125 µg: Healthy older adult received three injections, each consisting of 125 μg of GBS-NN and 125 μg of GBS NN2 bound to aluminium hydroxide.
  GBS-NN/NN2: GBS-NN/NN2 bound to alhydrogel as an adjuvant
- Healthy Older Adult : Placebo: Healthy older adult received three injections of placebo.
  Placebo: Normal Saline 0.9 %
- Obese and/or Diabetic Older Adult : GBS-NN/NN2 50 µg: Obese and/or diabetic older adults received three injections, each consisting of 50 μg of GBS-NN and 50 μg of GBS NN2 bound to aluminium hydroxide.
  GBS-NN/NN2: GBS-NN/NN2 bound to alhydrogel as an adjuvant
- Obese and/or Diabetic Older Adult : GBS-NN/NN2 125 µg: Obese and/or diabetic older adults received three injections, each consisting of 125 μg of GBS-NN and 125 μg of GBS NN2 bound to aluminium hydroxide.
  GBS-NN/NN2: GBS-NN/NN2 bound to alhydrogel as an adjuvant
- Obese and/or Diabetic Older Adult : Placebo: Obese and/or diabetic older adults received three injections of placebo.
  Placebo: Normal Saline 0.9 %
Period: Overall Study
Arm/Group | Healthy Older Adult : GBS-NN/NN2 50 µg | Healthy Older Adult : GBS-NN/NN2 125 µg | Healthy Older Adult : Placebo | Obese and/or Diabetic Older Adult : GBS-NN/NN2 50 µg | Obese and/or Diabetic Older Adult : GBS-NN/NN2 125 µg | Obese and/or Diabetic Older Adult : Placebo
Started | 24 | 24 | 12 | 12 | 12 | 6
Completed | 24 | 24 | 10 | 12 | 12 | 6
Not Completed | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Older Adult : GBS-NN/NN2 50 µg | Healthy Older Adult : GBS-NN/NN2 125 µg | Healthy Older Adult : Placebo | Obese and/or Diabetic Older Adult : GBS-NN/NN2 50 µg | Obese and/or Diabetic Older Adult : GBS-NN/NN2 125 µg | Obese and/or Diabetic Older Adult : Placebo | Total
Number analyzed (Participants) | 24 | 24 | 12 | 12 | 12 | 6 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (5.4) | 64.5 (5.5) | 65.8 (5.0) | 64.5 (6.0) | 65.4 (4.6) | 65.8 (1.3) | 65.1 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 4 | 7 | 8 | 4 | 45
  Male | 13 | 13 | 8 | 5 | 4 | 2 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 24 | 12 | 12 | 12 | 6 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 23 | 24 | 12 | 12 | 12 | 6 | 89
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 167.81 (10.50) | 168.98 (7.58) | 167.12 (7.85) | 171.88 (9.36) | 169.15 (11.67) | 172.00 (14.49) | 169.03 (9.65)
Weight [Mean (Standard Deviation); unit: Kg] | 70.98 (13.16) | 70.65 (7.45) | 68.88 (11.75) | 95.68 (12.54) | 95.38 (14.09) | 95.07 (11.91) | 78.76 (16.41)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.993 (2.537) | 24.808 (2.854) | 24.668 (3.856) | 32.262 (1.584) | 33.323 (3.340) | 32.437 (5.123) | 27.476 (4.772)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of the GBS-NN/NN2 Vaccine for 4 Weeks After Each Dose of Vaccine
Description: * Safety and tolerability as determined by the occurrence of Adverse Events (AEs) consisting of local and systemic reactogenicity within 7 days after vaccination
  * Unsolicited AEs, including adverse events of special interest (AESIs), Medically attended adverse events (MAAEs) and Serious adverse events (SAEs) within 28 days after each vaccination
  * AESIs, MAAEs, ARs/SARs leading to withdrawal from the study.
Time Frame: Up to 28 days after each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Older Adult : GBS-NN/NN2 50 µg | Healthy Older Adult : GBS-NN/NN2 125 µg | Healthy Older Adult : Placebo | Obese and/or Diabetic Older Adult : GBS-NN/NN2 50 µg | Obese and/or Diabetic Older Adult : GBS-NN/NN2 125 µg | Obese and/or Diabetic Older Adult : Placebo
Number analyzed (Participants) | 24 | 24 | 12 | 12 | 12 | 6
Participants
  Local Solicited AEs | 23 | 21 | 5 | 10 | 10 | 2
  Systemic Solicited AEs | 12 | 14 | 6 | 8 | 7 | 4
  Unsolicited AEs | 17 | 16 | 10 | 9 | 9 | 4
  AEs leading to withdrawal | 0 | 0 | 2 | 0 | 0 | 0

2. Secondary Outcome: Geometric Mean Antibody Concentration in μg/mL for Antibodies to the Four Individual Alps
Description: Geometric mean antibody concentration in μg/mL for antibodies to the four individual Alps (Alp 1, Alp2/3, Rib and AlpC) to evaluate IgG antibody response to the GBS-NN/NN2 vaccine at Day 197 (principal immunological endpoint).
Time Frame: Day 197
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Healthy Older Adult : GBS-NN/NN2 50 µg | Healthy Older Adult : GBS-NN/NN2 125 µg | Healthy Older Adult : Placebo | Obese and/or Diabetic Older Adult : GBS-NN/NN2 50 µg | Obese and/or Diabetic Older Adult : GBS-NN/NN2 125 µg | Obese and/or Diabetic Older Adult : Placebo
Number analyzed (Participants) | 24 | 24 | 10 | 12 | 12 | 6
μg/mL
  Anti-Alp1 | 13.14 [9.18 to 18.81] | 12.34 [9.62 to 15.83] | 0.08 [0.03 to 0.21] | 8.34 [4.45 to 15.62] | 14.17 [7.73 to 25.95] | 0.15 [0.06 to 0.35]
  Anti-Alp2/3 | 12.69 [9.26 to 17.39] | 17.39 [9.36 to 19.51] | 0.04 [0.02 to 0.08] | 10.90 [5.52 to 21.52] | 14.52 [8.92 to 23.65] | 0.09 [0.02 to 0.42]
  Anti-AlpC | 13.69 [9.82 to 19.09] | 11.28 [7.15 to 17.80] | 0.04 [0.02 to 0.11] | 6.64 [2.64 to 16.68] | 14.11 [5.05 to 39.44] | 0.10 [0.03 to 0.35]
  Anti-Rib | 4.76 [2.84 to 7.97] | 4.55 [2.78 to 7.46] | 0.04 [0.02 to 0.08] | 3.67 [1.82 to 7.39] | 4.59 [1.58 to 13.37] | 0.06 [0.02 to 0.16]

3. Secondary Outcome: Geometric Mean Fold Increase in Antibody Concentration for Antibodies to the Four Individual Alps
Description: Geometric mean fold increase in antibody concentration for antibodies to the four individual Alps (Alp 1, Alp2/3, Rib and AlpC) to evaluate IgG antibody responses induced by the three vaccine doses, on a 0-, 1- and 6-month regimen, in older adult participants 4 weeks after each vaccination.
Time Frame: 4 weeks after each vaccination (Days 29, 57 and 197)
Measure: Number (95% Confidence Interval); unit: Geometric mean fold ratio
Arm/Group | Healthy Older Adult : GBS-NN/NN2 50 µg | Healthy Older Adult : GBS-NN/NN2 125 µg | Healthy Older Adult : Placebo | Obese and/or Diabetic Older Adult : GBS-NN/NN2 50 µg | Obese and/or Diabetic Older Adult : GBS-NN/NN2 125 µg | Obese and/or Diabetic Older Adult : Placebo
Number analyzed (Participants) | 24 | 24 | 12 | 12 | 12 | 6
Geometric mean fold ratio
  Alp1 - Day 29 | 34.04 [18.65 to 62.13] | 24.99 [14.12 to 44.24] | 1.04 [0.98 to 1.10] | 21.27 [6.47 to 69.87] | 43.16 [17.67 to 105.44] | 0.78 [0.47 to 1.30]
  Alp1- Day 57 | 70.98 [44.71 to 112.67] | 39.71 [25.59 to 61.63] | 1.09 [0.99 to 1.19] | 32.86 [17.58 to 61.42] | 47.89 [25.05 to 91.56] | 0.84 [0.63 to 1.11]
  Alp1 - Day 197 | 124.30 [79.84 to 193.52] | 106.77 [69.83 to 163.23] | 0.85 [0.48 to 1.49] | 56.11 [29.99 to 104.99] | 114.75 [74.02 to 177.89] | 1.46 [0.45 to 4.77]
  Alp2/3 - Day 29 | 40.97 [27.11 to 61.92] | 50.32 [29.30 to 86.45] | 0.98 [0.90 to 1.07] | 20.17 [4.26 to 95.44] | 82.64 [30.33 to 225.14] | 0.66 [0.24 to 1.79]
  Alp2/3 - Day 57 | 72.60 [51.19 to 102.96] | 76.23 [51.23 to 113.42] | 1.03 [0.93 to 1.15] | 39.29 [16.20 to 95.28] | 84.82 [41.61 to 172.89] | 0.88 [0.74 to 1.05]
  Alp2/3 - Day 197 | 148.15 [103.14 to 212.79] | 204.85 [131.19 to 319.86] | 0.69 [0.37 to 1.28] | 89.51 [39.87 to 200.93] | 205.88 [102.76 to 412.50] | 1.09 [0.39 to 3.02]
  AlpC - Day 29 | 59.09 [36.75 to 95.01] | 31.75 [16.42 to 61.40] | 1.10 [1.02 to 1.17] | 29.37 [6.67 to 129.21] | 45.62 [16.18 to 128.63] | 0.63 [0.24 to 1.71]
  AlpC - Day 57 | 102.29 [65.31 to 160.21] | 38.89 [21.45 to 70.50] | 1.15 [1.04 to 1.28] | 40.66 [15.51 to 106.59] | 44.84 [20.39 to 98.61] | 0.87 [0.69 to 1.09]
  AlpC - Day 197 | 115.60 [76.71 to 174.19] | 114.30 [67.90 to 192.40] | 0.45 [0.26 to 0.77] | 60.42 [23.95 to 152.45] | 91.27 [43.68 to 190.72] | 0.95 [0.23 to 3.95]
  Rib - Day 29 | 18.56 [11.85 to 29.09] | 26.62 [14.61 to 48.53] | 1.03 [0.97 to 1.09] | 25.74 [8.03 to 82.57] | 20.95 [5.94 to 73.86] | 1.00 [0.90 to 1.10]
  Rib - Day 57 | 30.74 [20.83 to 45.37] | 34.87 [22.59 to 53.83] | 1.09 [1.00 to 1.18] | 36.74 [15.40 to 87.64] | 24.06 [9.96 to 58.09] | 1.10 [0.76 to 1.61]
  Rib - Day 197 | 47.74 [31.94 to 71.35] | 69.42 [42.27 to 114.01] | 0.68 [0.45 to 1.03] | 54.05 [25.53 to 114.40] | 37.74 [15.31 to 93.03] | 0.58 [0.26 to 1.27]

4. Secondary Outcome: Seroconversion Rate at Any Time Post Vaccination
Description: Seroconversion rate (proportion of participants with a 4-fold increase above baseline - pre dose concentration) at any time post vaccination to assess whether pre existing antibody levels affect the vaccine-induced antibody response.
Time Frame: Up to 6 months after last vaccination
Measure: Number; unit: participants
Arm/Group | Healthy Older Adult : GBS-NN/NN2 50 µg | Healthy Older Adult : GBS-NN/NN2 125 µg | Healthy Older Adult : Placebo | Obese and/or Diabetic Older Adult : GBS-NN/NN2 50 µg | Obese and/or Diabetic Older Adult : GBS-NN/NN2 125 µg | Obese and/or Diabetic Older Adult : Placebo
Number analyzed (Participants) | 24 | 24 | 12 | 12 | 12 | 6
participants
  Anti-Alp1 (µg/mL) - Day 29 | 22 | 21 | 0 | 9 | 11 | 0
  Anti-Alp1 - Day 57 | 23 | 24 | 0 | 12 | 12 | 0
  Anti-Alp1 - Day 169 | 23 | 24 | 0 | 11 | 12 | 1
  Anti-Alp1 - Day 197 | 24 | 24 | 0 | 12 | 12 | 1
  Anti-Alp1 - Day 365 | 23 | 24 | 0 | 12 | 12 | 1
  Anti-Alp2/3 - Day 29 | 24 | 23 | 0 | 7 | 11 | 0
  Anti-Alp2/3 - Day 57 | 24 | 24 | 0 | 12 | 12 | 0
  Anti-Alp2/3 - Day 169 | 24 | 24 | 0 | 11 | 12 | 1
  Anti-Alp2/3 - Day 197 | 24 | 24 | 0 | 12 | 12 | 1
  Anti-Alp2/3 - Day 365 | 24 | 24 | 0 | 12 | 12 | 0
  Anti-AlpC - Day 29 | 24 | 21 | 0 | 8 | 11 | 0
  Anti-AlpC - Day 57 | 24 | 24 | 0 | 11 | 12 | 0
  Anti-AlpC - Day 169 | 24 | 20 | 0 | 11 | 10 | 2
  Anti-AlpC - Day 197 | 24 | 24 | 0 | 12 | 12 | 2
  Anti-AlpC - Day 365 | 24 | 22 | 0 | 12 | 11 | 2
  Anti-Rib - Day 29 | 22 | 21 | 0 | 10 | 10 | 0
  Anti-Rib - Day 57 | 23 | 24 | 0 | 11 | 10 | 0
  Anti-Rib - Day 169 | 21 | 21 | 0 | 11 | 10 | 0
  Anti-Rib - Day 197 | 23 | 24 | 0 | 12 | 11 | 0
  Anti-Rib - Day 365 | 22 | 22 | 0 | 12 | 10 | 0

5. Secondary Outcome: Proportion of Participants Achieving Antibody Concentrations for Antibodies to the Four Individual Alps
Description: Proportion of participants achieving antibody concentrations for antibodies to the four individual Alps (Alp 1, Alp2/3, Rib and AlpC) above specific thresholds (>1, >2, >4, and >8 µg/mL) at Days 29, 57, 169, and 197, to evaluate the immune response up to 6 months following the third dose.
Time Frame: Up to day 197
Measure: Number; unit: participants
Arm/Group | Healthy Older Adult : GBS-NN/NN2 50 µg | Healthy Older Adult : GBS-NN/NN2 125 µg | Healthy Older Adult : Placebo | Obese and/or Diabetic Older Adult : GBS-NN/NN2 50 µg | Obese and/or Diabetic Older Adult : GBS-NN/NN2 125 µg | Obese and/or Diabetic Older Adult : Placebo
Number analyzed (Participants) | 24 | 24 | 12 | 12 | 12 | 6
participants
  Alp 1 >1 µg/mL - Day 29 | 19 | 19 | 0 | 8 | 10 | 0
  Alp 1 >1 µg/mL - Day 57 | 23 | 23 | 0 | 10 | 11 | 0
  Alp 1 >1 µg/mL - Day 169 | 21 | 20 | 0 | 9 | 9 | 0
  Alp 1 >1 µg/mL - Day 197 | 23 | 24 | 0 | 12 | 12 | 0
  Alp 1 >2 µg/mL - Day 29 | 16 | 16 | 0 | 7 | 10 | 0
  Alp 1 >2 µg/mL - Day 57 | 22 | 18 | 0 | 9 | 10 | 0
  Alp 1 >2 µg/mL - Day 169 | 18 | 14 | 0 | 7 | 7 | 0
  Alp 1 >2 µg/mL - Day 197 | 23 | 24 | 0 | 11 | 12 | 0
  Alp 1 >4 µg/mL - Day 29 | 13 | 11 | 0 | 7 | 8 | 0
  Alp 1 >4 µg/mL - Day 57 | 17 | 12 | 0 | 7 | 8 | 0
  Alp 1 >4 µg/mL - Day 169 | 12 | 7 | 0 | 4 | 6 | 0
  Alp 1 >4 µg/mL - Day 197 | 23 | 24 | 0 | 10 | 11 | 0
  Alp 1 >8 µg/mL - Day 29 | 8 | 5 | 0 | 4 | 5 | 0
  Alp 1 >8 µg/mL - Day 57 | 13 | 8 | 0 | 5 | 5 | 0
  Alp 1 >8 µg/mL - Day 169 | 8 | 2 | 0 | 1 | 2 | 0
  Alp 1 >8 µg/mL - Day 197 | 19 | 18 | 0 | 5 | 8 | 0
  Alp2/3 >1 µg/mL - Day 29 | 20 | 20 | 0 | 8 | 11 | 0
  Alp2/3 >1 µg/mL - Day 57 | 23 | 21 | 0 | 9 | 11 | 0
  Alp2/3 >1 µg/mL - Day 169 | 20 | 20 | 0 | 9 | 12 | 0
  Alp2/3 >1 µg/mL - Day 197 | 24 | 24 | 0 | 12 | 12 | 0
  Alp2/3 >2 µg/mL - Day 29 | 17 | 17 | 0 | 8 | 11 | 0
  Alp2/3 >2 µg/mL - Day 57 | 20 | 19 | 0 | 9 | 10 | 0
  Alp2/3 >2 µg/mL - Day 169 | 18 | 16 | 0 | 8 | 9 | 0
  Alp2/3 >2 µg/mL - Day 197 | 23 | 24 | 0 | 12 | 12 | 0
  Alp2/3 >4 µg/mL - Day 29 | 12 | 12 | 0 | 7 | 8 | 0
  Alp2/3 >4 µg/mL - Day 57 | 17 | 16 | 0 | 9 | 8 | 0
  Alp2/3 >4 µg/mL - Day 169 | 11 | 11 | 0 | 7 | 6 | 0
  Alp2/3 >4 µg/mL - Day 197 | 23 | 21 | 0 | 10 | 11 | 0
  Alp2/3 >8 µg/mL - Day 29 | 6 | 5 | 0 | 4 | 5 | 0
  Alp2/3 >8 µg/mL - Day 57 | 9 | 7 | 0 | 6 | 5 | 0
  Alp2/3 >8 µg/mL - Day 169 | 5 | 4 | 0 | 3 | 2 | 0
  Alp2/3 >8 µg/mL - Day 197 | 19 | 18 | 0 | 8 | 10 | 0
  Rib >1 µg/mL - Day 29 | 18 | 18 | 0 | 8 | 8 | 0
  Rib >1 µg/mL - Day 57 | 20 | 18 | 0 | 9 | 8 | 0
  Rib >1 µg/mL - Day 169 | 18 | 14 | 0 | 8 | 6 | 0
  Rib >1 µg/mL - Day 197 | 22 | 20 | 0 | 11 | 10 | 0
  Rib >2 µg/mL - Day 29 | 13 | 11 | 0 | 6 | 8 | 0
  Rib >2 µg/mL - Day 57 | 18 | 16 | 0 | 8 | 7 | 0
  Rib >2 µg/mL - Day 169 | 11 | 12 | 0 | 6 | 4 | 0
  Rib >2 µg/mL - Day 197 | 19 | 20 | 0 | 9 | 9 | 0
  Rib >4 µg/mL - Day 29 | 7 | 9 | 0 | 4 | 6 | 0
  Rib >4 µg/mL - Day 57 | 11 | 11 | 0 | 5 | 5 | 0
  Rib >4 µg/mL - Day 169 | 6 | 4 | 0 | 3 | 3 | 0
  Rib >4 µg/mL - Day 197 | 16 | 16 | 0 | 6 | 7 | 0
  Rib >8 µg/mL - Day 29 | 3 | 2 | 0 | 2 | 3 | 0
  Rib >8 µg/mL - Day 57 | 5 | 1 | 0 | 3 | 3 | 0
  Rib >8 µg/mL - Day 169 | 3 | 1 | 0 | 1 | 2 | 0
  Rib >8 µg/mL - Day 197 | 9 | 9 | 0 | 4 | 5 | 0
  AlpC >1 µg/mL - Day 29 | 22 | 17 | 0 | 8 | 9 | 0
  AlpC >1 µg/mL - Day 57 | 23 | 18 | 0 | 10 | 10 | 0
  AlpC >1 µg/mL - Day 169 | 22 | 19 | 0 | 9 | 9 | 0
  AlpC >1 µg/mL - Day 197 | 24 | 24 | 0 | 11 | 11 | 0
  AlpC >2 µg/mL - Day 29 | 21 | 15 | 0 | 7 | 9 | 0
  AlpC >2 µg/mL - Day 57 | 21 | 16 | 0 | 9 | 9 | 0
  AlpC >2 µg/mL - Day 169 | 21 | 18 | 0 | 6 | 8 | 0
  AlpC >2 µg/mL - Day 197 | 23 | 22 | 0 | 10 | 10 | 0
  AlpC >4 µg/mL - Day 29 | 15 | 12 | 0 | 6 | 8 | 0
  AlpC >4 µg/mL - Day 57 | 20 | 12 | 0 | 6 | 9 | 0
  AlpC >4 µg/mL - Day 169 | 15 | 10 | 0 | 4 | 6 | 0
  AlpC >4 µg/mL - Day 157 | 23 | 20 | 0 | 6 | 10 | 0
  AlpC >8 µg/mL - Day 29 | 11 | 7 | 0 | 5 | 7 | 0
  AlpC >8 µg/mL - Day 57 | 19 | 9 | 0 | 5 | 7 | 0
  AlpC >8 µg/mL - Day 169 | 5 | 5 | 0 | 3 | 5 | 0
  AlpC >8 µg/mL - Day 197 | 21 | 17 | 0 | 6 | 9 | 0

6. Secondary Outcome: Long-term Safety Profile of the GBS-NN/NN2 Vaccine Between Day 57 (28 Days Post Second Injection) to Day 168 and 6 Months Following the Third Dose (Safety Endpoint)
Description: * Proportion of participants with any SAE from between Day 57 (28 days post second injection) to Day 168 and 28 days after third vaccination (Day 197) up to Day 365.
  * Proportion of participants with MAAEs, AESIs, ARs/SARs requiring a medical consultation, and or leading to withdrawal from the study from 28 days after third vaccination (Day 197) up to Day 365.
Time Frame: Up to day 365
Measure: Number; unit: participants
Arm/Group | Healthy Older Adult : GBS-NN/NN2 50 µg | Healthy Older Adult : GBS-NN/NN2 125 µg | Healthy Older Adult : Placebo | Obese and/or Diabetic Older Adult : GBS-NN/NN2 50 µg | Obese and/or Diabetic Older Adult : GBS-NN/NN2 125 µg | Obese and/or Diabetic Older Adult : Placebo
Number analyzed (Participants) | 24 | 24 | 12 | 12 | 12 | 6
participants
  SAE from Day 57 to Day 168 | 0 | 0 | 1 | 0 | 0 | 0
  SAE from Day 197 to Day 365 | 0 | 1 | 1 | 0 | 0 | 0
  MAAEs from Day 197 up to Day 365 | 12 | 9 | 2 | 1 | 5 | 2
  AESIs from Day 197 up to Day 365 | 0 | 0 | 1 | 0 | 0 | 0
  ARs/SARs from Day 197 up to Day 365 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events were collected from Day 1 until Day 57 and from Day 162 to Day 197. From Day 58 to Day 16 and from Day 198 to Day 365, only MAAEs, AESIs, and SAEs were collected.
Arm/Group | Healthy Older Adult : GBS-NN/NN2 50 µg | Healthy Older Adult : GBS-NN/NN2 125 µg | Healthy Older Adult : Placebo | Obese and/or Diabetic Older Adult : GBS-NN/NN2 50 µg | Obese and/or Diabetic Older Adult : GBS-NN/NN2 125 µg | Obese and/or Diabetic Older Adult : Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/12 | 0/12 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/24 | 2/12 | 1/12 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 17/24 | 16/24 | 10/12 | 9/12 | 9/12 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Older Adult : GBS-NN/NN2 50 µg (N=24) | Healthy Older Adult : GBS-NN/NN2 125 µg (N=24) | Healthy Older Adult : Placebo (N=12) | Obese and/or Diabetic Older Adult : GBS-NN/NN2 50 µg (N=12) | Obese and/or Diabetic Older Adult : GBS-NN/NN2 125 µg (N=12) | Obese and/or Diabetic Older Adult : Placebo (N=6)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Older Adult : GBS-NN/NN2 50 µg (N=24) | Healthy Older Adult : GBS-NN/NN2 125 µg (N=24) | Healthy Older Adult : Placebo (N=12) | Obese and/or Diabetic Older Adult : GBS-NN/NN2 50 µg (N=12) | Obese and/or Diabetic Older Adult : GBS-NN/NN2 125 µg (N=12) | Obese and/or Diabetic Older Adult : Placebo (N=6)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Injection site warmth (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (5) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burnout syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT05782179/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT05782179/SAP_001.pdf